CLINICAL TRIAL: NCT01193569
Title: The SOS Study: A Study of Survival and Outcome After Stroke
Brief Title: A Study of Survival and Outcome After Stroke
Acronym: SOS
Status: Completed | Type: Observational
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP2818; CLP2818
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Standard of Care: Standard of Care for stroke except mechanical therapy

SUMMARY:
The objective of this study is to determine the natural history of acute ischemic stroke from large vessel thromboembolism in the brain. The target population is a stroke cohort with a known infarct volume who presents within 8 hours from symptom onset with a NIH Stroke Scale (NIHSS) score >10 who are eligible for mechanical thrombectomy but without receiving the treatment. Functional outcome as defined by the modified Rankin Scale (mRS) of all enrolled patients will be followed for 90 days after the index event.

DETAILED DESCRIPTION:
The objective of this observational study is to determine the natural history of acute ischemic stroke from large vessel thromboembolism in the brain. The target population is a stroke cohort with a known infarct volume who presents within 8 hours from symptom onset with a NIH Stroke Scale (NIHSS) score >10. Functional outcome as defined by the modified Rankin Scale (mRS) of all enrolled patients will be followed for 90 days after the index event. This is a prospective, single arm, multi-center trial. Up to 200 patients at up to 30 centers will be enrolled in the study. It is anticipated that up to 150 evaluable patients will be needed for analysis. The sample size estimate is based on the primary study functional outcome at 90 days as defined by a mRS of 0-2. Assuming that this observational study will have as outcome of 25% (37/150) mRS 0-2 at day 90, the expected two-sided exact binomial confidence interval is (18%, 32%). This sample size is adequate to estimate the mRS outcome of 0-2 at day 90 for the natural history of acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 85 years of age
* Evidence of proximal anterior circulation large vessel occlusion (TIMI 0-1/TICI 0-1)from CT Angiography. Target vessel occlusion may include the supra-clinoid segment of the ICA through the M1 segment of the MCA.
* Presented with symptoms consistent with acute ischemic stroke within 8 hours of symptom onset. Patients who presented within 3 hours must be ineligible or refractory to IV rtPA therapy.
* At time of enrollment, neurological deficit resulting in an NIH Stroke Scale (NIHSS) score > 10
* Known core infarct volume assessed by CTP, CTA or DWI scans

Exclusion Criteria:

* History of stroke in the past 3 months.
* Pre-existing neurological or psychiatric disease that could confound the study results such as a pre-stroke mRS score >1
* Known severe allergy to contrast media
* Uncontrolled hypertension (defined as systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg)
* CT evidence of the following conditions before enrollment:

  * Significant mass effect with midline shift
  * Evidence of intracranial hemorrhage
* Treated with endovascular therapy for acute stroke
* Life expectancy was thought to be less than 90 days prior to stroke due to non-stroke illness
* Participation in another clinical investigation that could confound the evaluation of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with symptoms of acute ischemic stroke within 8 hours from symptom onset and with an imaging-defined large cerebral vessel occlusion and a known infarct volume will be enrolled and followed for 90-days.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2010-09; Primary Completion 2016-12-22 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a modified Rankin score of 2 or less | 90 days after the procedure

SECONDARY OUTCOMES:
NIHSS score of 0-1 or a 10 or more points improvement | Discharge
All cause mortality | 90 days post-procedure
Incidents of symptomatic and asymptomatic intracranial hemorrhage | 90 days post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Iris Q Grunwald, MD, Principal Investigator — The John Radcliffe Hospital, Oxford, UK
Locations (1):
- Acute Vascular Imaging Centre, John Radcliffe Hospital, University of Oxford, Oxford, United Kingdom